CLINICAL TRIAL: NCT03179254
Title: Oral Hypoglycemic Agent Continuation Versus Interruption in Type 2 Diabetic Patients Undergoing Ambulatory Surgery
Brief Title: Type 2 Diabetes and Ambulatory Surgery Patients
Acronym: Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jin Meng, Medical Doctor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 032011-162
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hypoglycemic agent continue (Experimental): Metformin continue on the day of surgery
  Interventions: Drug: Metformin continue
- Oral hypoglycemic agent discontinue (Active Comparator): Metformin discontinue on the day of surgery
  Interventions: Drug: Metformin discontinue

INTERVENTIONS:
Drug: Metformin continue — Oral hypoglycemic agent continue on the day of ambulatory surgery
  Other Names: Metformin
  Arms: Oral hypoglycemic agent continue
Drug: Metformin discontinue — Oral hypoglycemic agent discontinue on the day of ambulatory surgery
  Other Names: Metformin
  Arms: Oral hypoglycemic agent discontinue

SUMMARY:
Patients scheduled to undergo ambulatory surgery are usually made non per os (NPO) at midnight on the day prior to surgery. In the case of patients with type 2 diabetic mellitus (DM) on treatment with oral hypoglycemic agent (OHA), patients are instructed to temporarily discontinue treatment on the day prior to surgery. This advice is based on the concern for intraoperative and postoperative hypoglycemia in this group of patients. Metformin , a dimethylbiguanide, is widely used as an oral antihyperglycemic drug in the long term treatment of type 2 DM. This instruction to withhold treatment may be imprudent given that metformin by virtue of its mechanism of action does not cause hypoglycemia. Another concern often cited as a reason to withhold metformin is the reported adverse effect of lactic acidosis. However, a recent metanalysis by the Cochrane group found no cases of fatal or nonfatal lactic acidosis in 70,490 patient-years of metformin use, or in 55,451 patient-years for those not on metformin. Furthermore, discontinuing OHA treatment can result in disruption of established glycemic control and intraoperative and postoperative hyperglycemia all of which can be deleterious to the patient.

We hypothesize that uninterrupted treatment with OHA in type 2 DM patients undergoing ambulatory surgery will not result in intraoperative and postoperative hypoglycemia (defined as blood glucose < 60mg/dl) compared to patients withholding OHA treatment on the day of surgery.

DETAILED DESCRIPTION:
Patients with established diagnosis of type 2 Diabetes Mellitus (DM) who are on OHA monotherapy or combination OHA and are scheduled to undergo ambulatory surgery will be identified. Informed consent will be obtained from 160 consecutive study participants. Patients will be randomized into 2 groups - OHA treatment on day of surgery (Metformin continue) (H1 group, n= 80) and patients not receiving OHA on day of surgery (OHA discontinue) (H0, n=80) as prescribed by their provider. All patients will be processed through the anesthesia preoperative clinic and instructions regarding preoperative medication handling will be provided to study participants by the investigator. The instructions will be reinforced by the clinic nursing staff in the usual fashion.

On the morning of the surgical procedure, the investigator will verify that medication administration instructions provided to the study participant was adhered to. The patient will be checked-in into the ambulatory surgery suite and usual surgical preparatory procedures followed. Pre-anesthesia capillary blood glucose measurement will be performed and recorded in the pre-surgical area.

Anesthesia will be induced and maintained in the usual fashion. Intraoperative capillary blood glucose levels will be checked and recorded.The investigator will ensure that glucose containing maintenance intravascular fluids are avoided throughout the anesthesia and surgery unless specifically indicated for treatment. All patients will be awakened and extubated at the end of surgery and transferred to the post anesthesia recovery (PAR) area as appropriate. Capillary blood glucose will be measured after arrival in the PAR. The capillary glucose tests obtained in this study is part of established and standard care and will be paid for by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years old
* Established diagnosis of type 2 diabetes mellitus
* Undergoing ambulatory surgery.
* Receiving OHA treatment for diabetes .

Exclusion Criteria:

* Treatment of insulin monotherapy
* Treatment with combination of oral hypoglycemic agents such as Thiazolidinediones-Repaglimide (Prandin), Rosiglitazone (Avandia), Pioglitazone (Actos).
* Renal Insufficiency with Serum Creatinine > 2mg/dl
* Decompensated congestive heart failure decompensated congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-08-26 (Actual)

PRIMARY OUTCOMES:
Postoperative blood glucose level | Within 1 hour arrival of the Postanesthesia Care Unit (PACU)
  Postoperative blood glucose level

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gasanova I, Meng J, Minhajuddin A, Melikman E, Alexander JC, Joshi GP. Preoperative Continuation Versus Interruption of Oral Hypoglycemics in Type 2 Diabetic Patients Undergoing Ambulatory Surgery: A Randomized Controlled Trial. Anesth Analg. 2018 Oct;127(4):e54-e56. doi: 10.1213/ANE.0000000000003675. PMID 30044293
- [Derived] Zerillo J, Agarwal P, Poeran J, Zubizarreta N, Poultsides G, Schwartz M, Memtsoudis S, Mazumdar M, DeMaria S Jr. Perioperative Management in Hepatic Resections: Comparative Effectiveness of Neuraxial Anesthesia and Disparity of Care Patterns. Anesth Analg. 2018 Oct;127(4):855-863. doi: 10.1213/ANE.0000000000003579. PMID 29933267